CLINICAL TRIAL: NCT06561321
Title: An Open-label, Phase II Study to Evaluate the Clinical Efficacy and Safety of Tapinarof for Adult Patients With Palmoplantar Keratoderma
Brief Title: Study to Evaluate the Safety and Efficacy of Tapinarof in Adults With Palmoplantar Keratoderma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Organon and Co (Industry)
Responsible Party: Principal Investigator, David Rosmarin, Chair, Department of Dermatology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21197
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Palmoplantar Keratoderma
Keywords: Dermatology
MeSH Terms: conditions — Keratoderma, Palmoplantar | interventions — tapinarof

STUDY DESIGN:
Intervention Model Description: The treatment duration will span 16 weeks.
  1. Following this 16-week period, participants who achieve disease clearance may discontinue the treatment. Patients who stop treatment at 16 weeks will be assessed for their sustained drug response, and their status of clearance will be followed at regularly scheduled visits up to 52 weeks.
  2. For those whose condition has not cleared, they will continue with the extension period with the treatment from 16 weeks until their disease becomes clear or until the conclusion of the study (52 weeks), whichever comes first.
  At the 52-week there will be a follow-up visit for all patients to monitor the response and check if they have maintained their response. As the drug already has a good safety profile and multiple assessments/outcome measures are being implemented, no additional follow-up is necessary but patients will be educated to come in for check-ups if any AEs persist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tapinarof Drug Treatment (Experimental): Subjects in this arm will apply Tapinarof 1% cream topically once daily for a 16-week open-label treatment period. Participants who achieve disease clearance after 16 weeks may discontinue treatment and will be monitored for sustained response up to 52 weeks. Those who do not achieve clearance will continue the treatment during an extension period for up to 36 additional weeks or until clearance is achieved, whichever comes first. Regular follow-up visits will assess the duration of disease clearance and monitor for any potential recurrence of keratoderma.
  Interventions: Drug: Tapinarof

INTERVENTIONS:
Drug: Tapinarof — Daily topical Tapinarof use will stop disease advancement and improve the quality of life in patients with palmoplantar keratoderma, through its AhR & NRF2 agonism properties.

SUMMARY:
The purpose of this study is to assess adults with palmoplantar keratoderma (thickening skin layer on palms and soles) who are treated with the study drug, tapinarof. This is a naturally occuring compound used for the treatment of psoriasis. This study is being done to find out how well and safe this drug is for stopping or treating keratoderma. This study aims to investigate the positive impacts of daily topical Tapinarof use in the improvement of Keratoderma. Clinical efficacy and safety profile of prescribing Tapinarof for this condition will be evaluated.

DETAILED DESCRIPTION:
This study aims to assess the benefits of the treatment. Should the treatment demonstrate benefits (as defined by the primary outcome measure) without any observed serious adverse events (SAEs), further clinical trials would be justified. If at least 2 out of 6 subjects benefits from the treatment (as defined by our primary outcome measure) and there are no SAEs, future clinical trials would be warranted. This initial data will determine whether it is worthwhile to proceed with a phase 2 trial, that will be both blinded and well-controlled.

The study is designed to gather preliminary experiences that can be used to design subsequent, well-controlled studies that are appropriately powered for statistical analysis. Currently, there is not enough experience with this medication in treating this specific condition, which is necessary to design successful randomized controlled trials (RCTs) for regulatory approval by the FDA. In dermatology, conducting studies in this manner is standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Ability to discern and provide written informed consent and voluntarily adhere to all of the protocol requirements
* Male or female subjects in their adult years (≥ 18 years of age), inclusive, from the time of providing written subject-investigator agreement.
* Confirmed clinical diagnosis of palmoplantar keratoderma.

Exclusion Criteria:

* Treatment with any of the following medications and therapies during the duration of the study*:

  * Topical corticosteroids
  * Keratolytic agents (eg, 6% salicylic acid, 70% propylene glycol, 30% water)
  * Topical retinoids
  * Topical vitamin D ointment (calcipotriol)
  * Oral retinoids (acitretin)

    * If on any of these then a washout period of at least 2 weeks will be enforced before the study begins. This washout period is meant to ensure that any effects or residues from previous treatments are minimized before starting the study.
* Prior exposure to Tapinarof treatment
* Known history or suspicion of hypersensitivity reactions, or contraindications to any or all components of the drug or drugs of similar properties.
* Currently participating in another clinical study for the same purpose.
* Potential or confirmed pregnancy: Individuals who are currently pregnant or have confirmed pregnancy at the time of screening will be excluded from participation in the study. This criterion aims to ensure the safety of participants and adhere to ethical considerations regarding the potential risks associated with the study interventions during pregnancy.
* Any other factors specifically not listed above but deemed patient unsuitable by the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) | Week 16 (Visit 4)
  To evaluate the treatment benefit of Tapinarof applied topically to patients affected with palmoplantar keratoderma.
  Either an overall change in the PGA score to 0 (clear) or 1 (almost clear) or a decrease from baseline of at least 2 points. Higher scores indicate a worse outcome.
  Title: PHYSICIAN GLOBAL ASSESSMENT Minimum value: 0 Maximum value: 5

SECONDARY OUTCOMES:
Treatment Emergent Adverse Event (TEAEs) | through study completion, 52 weeks
  To assess the safety of Tapinarof applied topically to patients affected with palmoplantar keratoderma.
  Frequency and severity of treatment emergent adverse events (TAEs).
Skin assessment every visit | through study completion, 52 weeks
  To assess additional measures of efficacy of Tapinarof applied topically to patients affected with palmoplantar keratoderma, through qualitative analysis done by the investigator.
  Skin assessment of the affected areas, palms and/or soles, that are being managed with topical Tapinarof.
Skin pictures at baseline to 52 weeks | through study completion, 52 weeks
  To assess additional measures of efficacy of Tapinarof applied topically to patients affected with palmoplantar keratoderma, through qualitative analysis done by the investigator.
  To identify and note any visible differences due to the application of Tapinarof, throughout the treatment phase from baseline, 4 weeks, end of primary endpoint and lastly at the end of the monitoring phase at 52 weeks.
Patient Global Assessment (PtGA) | through study completion, 52 weeks
  To assess additional measures of efficacy of Tapinarof applied topically to patients affected with palmoplantar keratoderma, through qualitative analysis done by the patient.
  Note any patient reported outcomes and patient satisfaction of the treatment through a standardized Patient Global Assessment (PtGA) questionnaire. Higher scores indicate a worse outcome.
  Title: PATIENT GLOBAL ASSESSMENT Minimum value: 0 Maximum value: 5
Dermatology Life Quality Index (DLQI) | through study completion, 52 weeks
  To assess additional measures of efficacy of Tapinarof applied topically to patients affected with palmoplantar keratoderma, through qualitative analysis done by the patient. Done to monitor patient's observation and impact of Tapinarof use to their quality of life. Higher scores indicate a worse outcome.
  Title: DERMATOLOGY LIFE QUALITY INDEX Minimum value: 0 Maximum value: 30

CONTACTS AND LOCATIONS:
Overall Officials: David Rosmarin, MD, Principal Investigator — Dermatology
Locations (1):
- Indiana University Department of Dermatology, Indianapolis, Indiana, United States

REFERENCES:
- See also: Kerns ML;Hakim JM;Lu RG;Guo Y;Berroth A;Kaspar RL;Coulombe PA; (n.d.). Oxidative stress and dysfunctional Nrf2 underlie Pachyonychia Congenita phenotypes. The Journal of clinical investigation — https://pubmed.ncbi.nlm.nih.gov/27183391/
- See also: Keam, S. J. (2022, August 17). Tapinarof Cream 1%: First approval - drugs. SpringerLink — http://link.springer.com/article/10.1007/s40265-022-01748-6